CLINICAL TRIAL: NCT00782301
Title: A Multicenter, Randomized, Open, Comparative Trial Of Maraviroc Versus Etravirine Each In Combination With Darunavir/Ritonavir And Raltegravir For The Treatment Of Antiretroviral-Experienced HIV-1 Subjects Co-Infected With Hepatitis C And/Or Hepatitis B
Brief Title: Maraviroc Versus Etravirine In Combination With Antiretroviral Therapy In Drug Experienced HIV And Hepatitis Co-Infected Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4001080
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Hepatitis B; Human Immunodeficiency Virus; Hepatitis C, Chronic
Keywords: HIV and Hepatitis co-infection
MeSH Terms: conditions — Hepatitis B; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic | interventions — Maraviroc; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maraviroc (Active Comparator)
  Interventions: Drug: maraviroc
- Etravirine (Active Comparator)
  Interventions: Drug: etravirine

INTERVENTIONS:
Drug: maraviroc — maraviroc 150 mg. p.o. b.i.d., darunavir 600 mg. p.o. b.i.d., ritonavir 100 mg. p.o. b.i.d., raltegravir 400 mg. p.o. b.i.d.
  Other Names: Selzentry
  Arms: Maraviroc
Drug: etravirine — etravirine 200 mg. p.o. b.i.d., darunavir 600 mg. p.o. b.i.d., ritonavir 100 mg. p.o. b.i.d., raltegravir 400 mg. p.o. b.i.d.
  Arms: Etravirine

SUMMARY:
Confirm the safety of maraviroc when used as a component of combination antiretroviral therapy in HIV and Hepatitis co-infected patients.

ELIGIBILITY:
Inclusion Criteria:

HIV-1 RNA viral load of ≥1000 copies/mL at the screening visit. Detectable HCV RNA levels or Hepatitis B surface antigen (HBsAg) positive. Previous antiretroviral treatment experience with at least 2 antiretroviral drug classes for ≥3 months.

Documented resistance to an NNRTI as well as documented resistance to another antiretroviral agent.

CCR5 tropic virus detected by the TrofileTM assay.

Exclusion Criteria:

Suspected or documented active, untreated HIV-1 related Opportunistic Infection (OI) or other condition requiring acute therapy at the time of randomization (subjects on a stable (>1 month) secondary OI prophylaxis regimen are eligible for the study; subjects on a primary OI prophylaxis regimen of any duration are also eligible for the study).

Prior treatment with darunavir/ritonavir, raltegravir, or another integrase inhibitor, etravirine, maraviroc or another CCR5 inhibitor for more than 14 days at any time.

Subjects receiving treatment for chronic Hepatitis or the expected need to initiate HCV treatment within 48 weeks of randomization. (Subjects who were previously treated for Hepatitis C are eligible for the study).

AST and/or ALT greater than 5 times the upper limit of normal (ACTG Grade 3).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with Grade 3 and Grade 4 ALT test abnormalities associated with a change from baseline ALT ≥100 IU/L through Week 48. | 48 weeks

SECONDARY OUTCOMES:
Percentage of HCV treated subjects with Grade 3 and Grade 4 ALT test abnormalities associated with a change from baseline ALT ≥100 IU/L through 96. | 48 weeks
Time to development of Grade 3 and Grade 4 ALT test abnormalities associated with a change from baseline ALT ≥100 IU/L. | 96 weeks
Percentage of subjects with Hy's law abnormalities through Week 48. | 48 weeks
Percentage of HCV treated subjects with Hy's law abnormalities through Week 96. | 96 weeks
Change from baseline in mean Hepatitis C viral load through Week 48 | 48 weeks
Undetectable HCV viral load 24 weeks after stopping HCV treatment. | 240 weeks
Percentage of subjects with HIV-1 RNA levels <48 copies/mL at Week 48. | 48 weeks
Change from baseline in CD4+ cell count at Week 48. | 48 weeks
Change from baseline in mean hepatitis B DNA through Week 48 | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (13):
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, Wilton Manors, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Mount Vernon, New York
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Conroe, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Stafford, Texas
- Canada (2):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Toronto, Ontario
- Pfizer Investigational Site, Bydgoszcz, Poland

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001080&StudyName=Maraviroc%20Versus%20Etravirine%20In%20Combination%20With%20Antiretroviral%20Therapy%20In%20Drug%20Experienced%20HIV%20And%20Hepatitis%20Co-Infected%20Patients